CLINICAL TRIAL: NCT04939025
Title: Multi-interventional Program to Reduce Chronic Ileoanal Pouch Leaks in UC
Acronym: MIRACLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 271078
Record Dates: First submitted 2021-06-23; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
Keywords: ileoanal pouch, IPAA, pouch, ulcerative colitis, leak
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: The MIRACLE study is an international multicenter clinical effectiveness study, whereby the current local practice (control cohort) will be evaluated, and subsequently compared to the results after implementation of the multi-interventional program (intervention cohort).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historic cohort (No Intervention)
- Multi-interventional program cohort (Other)
  Interventions: Procedure: Multi-interventional program

INTERVENTIONS:
Procedure: Multi-interventional program — 1. Preoperative oral antibiotics and antibiotic enema of the rectal stump prior to the surgery
  2. Routine and tailored lengthening measures of the mesentery
  3. Intraoperative control of pouch vascularization using ICG
  4. Early diagnosis and active assessment of the integrity of the anastomosis.
     1. Routine CRP-measurements at day 4 and 6 (after removal pouch catheter) in the non-diverted pouches with CT-scan with rectal contrast if any suspicion on a leak (elevated or rise in CRP. symptoms).
     2. Routine CRP-measurements at day 4 in the diverted pouches with endoscopy 10-14 days after pouch creation.
  5. Endosponge vacuum assisted closure (EVAC) of the anastomotic defect aiming to close the defect within 10-14 days after diagnosis.
  6. MRI assessment of the pouch after stoma closure preferably at one year to rule out chronic sepsis mimicking pouchitis or Crohn's disease.
  Arms: Multi-interventional program cohort

SUMMARY:
The objective of this quality improvement project is to increase the one year anastomotic integrity rate in patients having had completion proctectomy and pouch reconstruction for Ulcerative Colitis by the routine and quality controlled implementation of a multi-interventional program thereby improving long-term pouch function and survival.

DETAILED DESCRIPTION:
Ulcerative colitis is an inflammatory bowel disorder that affects predominantly young patients interfering with their social, family and professional life's (Ungaro, Mehandru, Allen, Peyrin-Biroulet, & Colombel, 2017). When the disease is moderate to severe, it is difficult to control medically even in the era of the biologic treatment. Colectomy rates are reported to be as high as 50% after 5 years in patients admitted with a severe exacerbation (Duijvis et al., 2016; Thorne et al., 2016). In a modified two (colectomy first followed by completion proctectomy and pouch) or three stage procedure (colectomy first followed by completion proctectomy and pouch with diverting ileostomy, finally stoma closure) a proctocolectomy is done and continuity can be restored with a ileoanal pouch (Sahami, Buskens, et al., 2016; Zittan et al., 2016). These are the preferred options for the majority of our patients. Alternatives are proctocolectomy with definitive end-ileostomy or a continent ileostomy.

Quality of life of patients with pouches depends predominantly on proper function of the pouch. Inadequate function and long term pouch failure are determined by the occurrence of chronic anastomotic leaks, chronic pouchitis and a delayed diagnosis of Crohn's disease in and around the pouch (Lightner et al., 2017). The latter two diagnoses, Crohn's disease and chronic pouchitis are in an important number in fact misdiagnosed chronic leaks (Garrett et al., 2009; van der Ploeg, Maeda, Faiz, Hart, & Clark, 2017). Long-term pouch failure rates (pouch excision or secondary diversion of the pouch) add up to more than 1 out of 10 at 10 years (Ikeuchi et al., 2018; Lightner et al., 2017; Mark-Christensen et al., 2018). These data represent the results of expert centers, so real life data are probably worse. Chronic leaks are late sequalae leaking anastomosis which has been inadequately treated; misdiagnosed or diagnosed too late to treat successfully.

Although many centers publish more favorable figures, the true rate of anastomotic leakage of ileoanal pouches probably varies from 10-20% (Sahami, Bartels, et al., 2016; Sossenheimer et al., 2019; Widmar et al., 2019). There is an important underreporting of the leaks. If the pouch is diverted, the leak will only become apparent prior to ileostomy closure when the anastomosis is tested. Even testing the anastomosis is not 100% accurate accounting for a number of misdiagnosed leaks. These misdiagnosed and delayed diagnosed leaks are generally not included in series reporting short term results (Santorelli, Hollingshead, & Clark, 2018; Sossenheimer et al., 2019; Widmar et al., 2019).

For all these reasons it is of great importance to prevent anastomotic leakage when creating a ileoanal pouch and if it happens, to solve the problem as soon as possible.

Numerous risk factors have been identified for anastomotic leakage. The most important factors are tension on the anastomosis, inadequate vascularization of the pouch, an unfavorable microbiome and the use of immunosuppressive drugs (steroids, immunomodulators, biologic treatments). By staging the restorative proctocolectomy, the negative impact of immunosuppressive drugs on anastomotic healing are avoided because at the time of the pouch creation the drugs are weaned for a long period. Other factors including anastomotic technique and anastomotic perfusion are modifiable surgical factors. A more recently described pathophysiological mechanism relates to the intestinal microbiome (Alverdy, Hyoju, Weigerinck, & Gilbert, 2017). Apparently, this holds true for small bowel surgery as well (Lesalnieks, Hoene, Bittermann, Schlitt, & Hackl, 2018).

Proper management of a leak comprises early diagnosis and immediate and adequate management. Sequential CRP measurement and early investigation of the integrity of the anastomosis are key for early diagnosis, particularly in a diverted anastomosis which might not be symptomatic (Adamina et al., 2015; Warschkow et al., 2012).

The current management of the leak usually involves a diverting ileostomy, if not performed primarily, in combination with passive drainage of the abscess cavity via transanal or transcutaneous route. This approach showed to be relatively ineffective leading to a pouch failure rate of 20%, and if resolved to a worse pouch function (Garrett et al., 2009; Lightner et al., 2017).

Endosponge vacuum assisted closure (EVAC) of the anastomotic leak on the contrary showed to have a very high success rate and to prevent long-term pouch dysfunction and failure (Bemelman & Baron, 2018; Gardenbroek et al., 2015; Verlaan et al., 2011; Weidenhagen, Gruetzner, Wiecken, Spelsberg, & Jauch, 2008).

There is minimal risk to patients as there is no introduction of a novel technique, rather this study is an amalgamation of published improvements in pouch surgery pre, intra and post-operatively to reduce the leak rate at one year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ulcerative Colitis
* Diagnosis of Crohn's disease limited to the colon without any history of perianal disease
* Modified two or three stage restorative proctocolectomy
* Age above 18
* Able to fill in questionnaires in local language and to come to out-patient-clinic visits;

Exclusion Criteria:

* Known allergy to ICG, or iodide allergy.
* Pregnancy
* Redo pouch operation
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Leak rate | 1 year
  Anastomotic integrity at one year postoperatively defined as the absence of presacral collections, anastomotic fistula and severe anastomotic stricture (not amenable for digital dilatation by rectal exam).

SECONDARY OUTCOMES:
Cumulative anastomotic dehiscence rate | 18 month
  Anastomotic insufficiency at 30 days, 6 months and 12 months defined as contrast extravasation and/or presacral perianastomotic fluid collections on CT scan or Anastomotic dehiscence at endoscopy.
QOL | 3,6,12 and 18 months
  Quality of life and functional outcomes preoperatively and then 3, 6, 12 and 18 months post-operatively.
Protocol compliance | 18 month
  Protocol compliance to any intervention
ICG | Operative
  Change in management due to ICG
CRP | 30 days
  Diagnostic accuracy of CRP for anastomotic leakage
EVAC | 18 month
  Efficacy of EVAC with early transanal closure of the anastomotic defect
Stoma rate | 18 month
  Permanent stoma rate at 18 months
Temporary ileostomy rate and duration | 18 month
  Temporary stoma rate and stoma duration at 18 months
Complications | 1 year
  Operative and post-operative complications within 30 days and 12 months (cumulative) of operation (using the Clavien-Dindo classification of surgical complications)
Death | 1 year
  Death
Hospital stay | 1 year
  Hospital stay and total hospital stay at one year
Reintervention rate | 18 month
  Reintervention rate
Readmission | 18 month
  Overall and stoma-related readmission
Cost analysis of EVAC | 18 month
  Cost analysis of anastomotic leakage and EVAC therapy